CLINICAL TRIAL: NCT02222285
Title: An Exploratory, Double-Blind, Placebo-Controlled Study of the Medical Food Vayarin in Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Vayarin_005
Record Dates: First submitted 2014-08-12; First posted 2014-08-21 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2017-01

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 3: placebo/placebo (Placebo Comparator): Placebo/placebo consists of placebo for 7 weeks followed by 7 weeks of placebo treatment
  Interventions: Other: Placebo
- Sequence 2: placebo/ Treatment (Active Comparator): Sequence 2: placebo/ Treatment , consists of placebo for 7 weeks followed by 7 weeks of treatment with Vayarin_005
  Interventions: Other: Medical Food : Vayarin_005; Other: Placebo
- Sequence one: Treatment/Treatment (Active Comparator): Treatment/Treatment- consists of PS_005 for 7 weeks followed by 7 weeks of additional treatment with Vayarin_005
  Interventions: Other: Medical Food : Vayarin_005

INTERVENTIONS:
Other: Medical Food : Vayarin_005
  Arms: Sequence 2: placebo/ Treatment; Sequence one: Treatment/Treatment
Other: Placebo
  Other Names: Cellulose
  Arms: Sequence 2: placebo/ Treatment; Sequence 3: placebo/placebo

SUMMARY:
The primary study objective is to evaluate the efficacy of Vayarin_005 on ASD related symptoms in children.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ages 6-17 inclusive
2. Must have a valid diagnosis of autism spectrum disorder via a clinical review of the DSM-IV, confirmed by Autism Diagnostic Observation Schedule (ADOS)
3. Clinical Global Impression Scale of Severity of Illness for Pervasive Developmental Disorders (CGI-S-PDD) rating of 4 or higher (moderately ill or worse)
4. IQ >50 evaluated by KBIT-2 or Stanford Binet Fifth Edition
5. Able, and likely to fully comply with the study procedures and instructions
6. Subjects with mood, anxiety, or disruptive behavior disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.
7. Have normal physical examination and laboratory test results at screening. If abnormal, the finding(s) must be deemed clinically insignificant by the study Clinician.
8. Parents or legal guardian must be able to read, write and speak English
9. Parents or legal guardian have given written informed consent to participate in the study

Exclusion Criteria:

1. The subject is significantly underweight under the 5th percentile or obese above the 95th percentile
2. Clinically significant systemic illness including hepatic, renal, gastroenterological, metabolic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease, as determined by the study clinician.
3. Patients with any primary psychiatric diagnosis other than autism at screening or a known genetic syndrome(s) that cause autism.
4. Suspected or established CNS injury
5. Change in dosage of psychiatric pharmacotherapy or other medications that have central nervous system effects or that affect performance 4 weeks before study initiation and throughout the study phase
6. Use of alpha-agonists, or ADHD medications 4 weeks prior to study initiation and throughout the study
7. Use of dietary supplements, 60 days before study initiation and throughout the study
8. Change in educational/behavioral interventions within one month prior to participation or during the study
9. A known comorbid psychiatric diagnoses of bipolar I disorder, suicidality, or substantial psychotic disorder.
10. Subject who has participated in another clinical trial within 30 days of screening for this trial and/or any experimental treatment for this population
11. Current history of physical, sexual, or emotional abuse
12. History of alcohol or substance abuse as defined by DSM-IV criteria
13. Consumption of >250 mg/day of caffeine
14. History of allergic reactions or sensitivity to marine products and soy
15. Has any illness which may jeopardize the participants' health or limit their successful trial completion.
16. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient safety

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist will be used to asses Autism spectrum symptoms | over 14 weeks
  A significant reduction from baseline to endpoint on the Aberrant Behavior Checklist (ABC) compared to patients administered placebo

SECONDARY OUTCOMES:
Clinical Global Impression of Severity assesment | over 14 weeks
Clinical Global Impression of Improvement assesment | over 14 weeks
Conners Rating Scale questionnaire | over 14 weeks
Behavior Rating Inventory of Executive function | over 14 weeks
Child Health Questionnaire | over 14 weeks
Caregiver Strain Questionnaire | over 14 weeks
Adverse events monitoring | over 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, M.D., Principal Investigator — Spectrum Neuroscience and Treatment Institute
Locations (2):
- United States (2):
  - Institute of Neurology and Neurosurgery at St. Barnabas, Livingston, New Jersey
  - Spectrum Neuroscience and Treatment Institute, New York, New York